CLINICAL TRIAL: NCT06257316
Title: A Study on the Appropriate Dosage of Vasopressors to Maintain Adequate Cerebral Blood Flow During Surgery and Anesthesia in Neonates and Infants
Brief Title: Appropriate Dosage of Vasopressor in Neonates and Infants
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2312-009-1489
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hypotension; Neonatal Hypotension; Intraoperative Complications
MeSH Terms: conditions — Hypotension; Intraoperative Complications | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0.1mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml
- 0.2mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml
- 0.3mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, and 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml
- 0.5mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, and 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml
- 1.0mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, and 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml
- 1.2mg/kg of ephedrine (Active Comparator): If the mean arterial pressure decreases by more than 20% from baseline after induction of anesthesia and infusion of fluids until the start of surgery, a randomized dose of ephedrine will be administered.
  Six single doses were evaluated using six cohorts (N=20 per cohort). Subjects received single doses of ephedrine intravenously: 0.1, 0.2, 0.3, 0.5, 1.0, and 1.2 mg/kg.
  Initially, 3 cohorts received the study drug at a given dose, after assessing the safety of ephedrine by the Korean Ministry of Food and Drug Safety, the additional 60 subjects in 3 cohorts received the study drug.
  Interventions: Drug: EPHEDrine Hydrochloride 5 mg/ml

INTERVENTIONS:
Drug: EPHEDrine Hydrochloride 5 mg/ml — In the present study, the expected rate of recovery of the internal carotid artery according to the dose of the inotropic agent was similar to that in a previous study in which the fraction maintaining mean arterial pressure within 80% of baseline by dose of inotropic agent was 0.9% for the ephedrine 0.1, 0.6, 0.8, 1. 0, 1.2, and 1.4 doses (mg/kg) were 9.9%, 21%, 41%, 47%, 65.5%, and 40%, respectively (Br J Anaesth. 2023 May;130(5):603-610), and it was assumed that the rate of internal carotid artery recovery by inotrope dose would be 90% of that result.
  The study will randomize to dose in six cohorts and will include dose group and cohort variables in a logistic regression model to assess the trend between inotropic dose and rate of carotid revascularization after correcting for cohort effects on the outcome variable.

SUMMARY:
In this study, the investigators will evaluate cerebral blood flow before and after drug infusion using ultrasound to suggest blood pressure criteria and dosage of ephedrine, a vasopressor, to maintain adequate cerebral blood flow in neonates and infants undergoing surgery and anesthesia.

DETAILED DESCRIPTION:
Improvements in surgical techniques and perioperative care in the neonate have resulted in a significant improvement in survival rates, with the mortality rate for neonatal noncardiac surgery being less than 5% in 2013, compared to 72% in 1947. As survival rates have improved, the question of long-term prognosis, especially concerning delayed cranial nerve development and subsequent quality of life, has emerged. In 48% of full-term infants undergoing non-cardiac surgery in the neonatal period for major congenital conditions (diaphragmatic hernia, esophageal atresia, abdominal wall defects, congenital megacolon, etc.) and 75% of preterm infants, brain damage is identified on post-operative brain MRI, and developmental testing reveals cognitive impairment in 3-56% and motor impairment in 0-77%.

motor disorders in 3-56% and 0-77%. Cognitive and motor deficits are known to occur in 45% of patients undergoing non-cardiac surgery for congenital conditions, excluding neurodevelopmental disorders caused by the concomitant congenital genetic disease itself.

Cerebral perfusion is regulated by arterial baroreflex, cerebral blood flow autoregulation, and flow metabolism, which are immature in the neonate and are lost under general anesthesia. This can lead to intraoperative changes in blood pressure, carbon dioxide concentration, intraventricular hemorrhage, and lateral ventricular hemorrhagic infarction, which can cause brain damage.

According to the Anaesthesia Practice in Children Observational Trial study, 32% of children undergoing general anesthesia and surgery develop hypotension that requires inotropes. The goal of maintaining arterial blood pressure at a constant level in infants during surgery is to maintain blood flow to vital organs, including the brain. However, there is a lack of evidence on what blood pressure should be maintained to maintain adequate cerebral perfusion in infants and how much hypotension is acceptable. The current definition of normal blood pressure in infants is based on birth weight and gestational age. For example, if the gestational age is 36 weeks, the recommendation is to maintain a mean arterial pressure of 36 mm Hg or higher. However, studies have shown that mean arterial pressure below this level does not affect prognosis as long as adequate perfusion is maintained. Furthermore, raising blood pressure to maintain normotension based on gestational age may lead to intraventricular hemorrhage. A recent study was published to determine the appropriate dose of ephedrine in infants with intraoperative hypotension and found that a higher dose (1.2 mg/kg) than the adult dose (0.1 mg/kg) was required to raise blood pressure, but the study was limited by the lack of confirmation of how raising blood pressure changes cerebral blood flow. Therefore, in this study, the investigators aimed to determine the changes in cerebral blood flow according to the dose of ephedrine infusion in neonates and infants as measured by the changes in blood flow in the internal carotid artery using transcranial ultrasound and to suggest blood pressure standards and ephedrine dosage for maintaining adequate cerebral blood flow in neonates and infants.

ELIGIBILITY:
Inclusion Criteria:

* Newborns and infants under 2 years of age undergoing surgery under general anesthesia at Seoul National University Hospital

Exclusion Criteria:

* Premature infants with a gestational age of less than 37 weeks
* Children with a history of brain disease (hydrocephalus, brain tumor, etc.)
* Patients with a history of hypoxic/ischemic brain injury
* Children with fused fontanels
* Children with uncorrected congenital cardiac malformations such as patent ductus arteriosus
* Patients with hypersensitivity to ephedrine and its components
* Patients with hypertension
* Patients with thyrotoxicosis
* Patients with renal impairment and those taking thyroid medication
* Glaucoma patients
* Diabetic patients
* Patients with prostatic hyperplasia
* Patients with chromophobe cell tumors
* Patients taking or within 2 weeks of discontinuing monoamine oxidase inhibitors
* Patients with ischemic heart disease
* Patients receiving foxglove preparations
* Patients with cardiac disease
* Patients receiving inotropic agents and those with abnormal baseline blood pressure
* Those who are taking or need to take concomitant contraindicated medications
* Those who require halogenated anesthetics such as chloroform, cyclopropane, and halothane because concomitant administration may cause ventricular arrhythmias.
* Those who are expected to require these agents because they may cause arrhythmias or cardiac arrest when coadministered with catecholamines such as epinephrine and isoproterenol.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Recovery of cerebral blood flow within 10 minutes | within 10 minutes after ephedrine injection
  Whether at least one of the peak systolic velocity, end diastolic velocity, or velocity time integral of the internal carotid blood flow recovers to at least 80% of the baseline value within 10 minutes of the bolus injection.

SECONDARY OUTCOMES:
Recovery of cerebral blood flow within 2 minutes | within 2 minutes after ephedrine injection
  Whether at least one of the peak systolic velocity, end diastolic velocity, or velocity time integral of the internal carotid blood flow recovers to at least 80% of the baseline value within 2 minutes of the bolus injection.
Recovery of cerebral blood flow within 5 minutes | within 5 minutes after ephedrine injection
  Whether at least one of the peak systolic velocity, end diastolic velocity, or velocity time integral of the internal carotid blood flow recovers to at least 80% of the baseline value within 5 minutes of the bolus injection.
Recovery of mean arterial pressure within 10 minutes | within 10 minutes after ephedrine injection
  Whether the mean arterial pressure recovers to at least 80% of the baseline value within 10 minutes of the bolus injection.
Additional durg dose | within 10 minutes after ephedrine injection
  Type and dose of additional inotropes administered if mean arterial pressure does not return to at least 80% of baseline within 10 minutes of ephedrine injection.
electroencephalogram | from the induction of anesthesia to initiation of surgery
  Hemodynamic changes and their relationship to changes in cerebral oxygen saturation and electroencephalogram
cerebral oxygen saturation | from the induction of anesthesia to initiation of surgery
  Hemodynamic changes and their relationship to changes in cerebral oxygen saturation and electroencephalogram
fluid responsiveness | from the induction of anesthesia to initiation of surgery
  Determine if the presence of fluid responsiveness affects changes in cerebral blood flow induced by ephedrine injection

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Hee Kim, M.D., Ph.D., Study Chair — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No